CLINICAL TRIAL: NCT07227116
Title: ESCALATE: Evaluating the Status of Complex Aneuploidy to Locate Additional Transferrable Embryos
Brief Title: Evaluating the Status of Complex Aneuploidy to Locate Additional Transferrable Embryos
Acronym: ESCALATE
Status: Recruiting | Type: Observational
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Principal Investigator, Benjamin Harris, MD, Shady Grove Fertility Reproductive Science Center
Other Study IDs: 20250101
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Complex Aneuploidy; Chaotic Aneuploidy
Keywords: Chaotic, Complex, Aneuploidies, Embryos
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA will be retained by the testing laboratory for quality control and confirmatory testing under IRB-approved protocols. No identifiable genetic material will be stored or used for future research beyond this study without additional consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Aneuploidy Embryos: Embryos identified by PGT-A as having multiple chromosomal aneuploidies. DNA from trophectoderm re-biopsy samples will be retained by the testing laboratory for confirmatory analysis and quality control under IRB-approved protocols.

SUMMARY:
This study aims to evaluate the reproductive potential of embryos classified as "complex aneuploid" (involving three or more abnormal chromosomes) or "chaotic" (six or more abnormal chromosomes) through preimplantation genetic testing for aneuploidy (PGT-A). Specifically, we seek to determine whether embryos initially reported as having multiple chromosomal abnormalities might still have the potential for normal chromosomal composition, the opportunity for transfer, and ultimately, the potential to achieve a live birth through re-biopsy and reanalysis.

Key Information:

This portion of the study seeks your consent for the re-biopsy and genetic reanalysis of the embryos only. It does not yet include consent for potential future transfer.

Participation remains completely voluntary, and your decision will not affect your current or future care.

We deeply appreciate your support and commitment to advancing fertility research.

DETAILED DESCRIPTION:
Recently, the term "chaotic" has come into the PGT-A reporting lexicon, defined (perhaps arbitrarily) as 6 or more aneuploidies detected. Complex aneuploidy refers to embryos with multiple chromosomal aneuploidies. In one large study, complex aneuploidy at the cleavage stage was found in 41% of embryos overall, 29% of embryos in women 27-37 years old, and 45% of embryos in women 38-45 years old. By the blastocyst stage, only 10% of all embryos were complex aneuploid, with 13.7% of embryos in women aged 38-47 years compared to 4.5% in women aged 27-37 years demonstrating complex aneuploidy. Multiple aneuploidies were also detected in a retrospective study of 1502 spontaneous abortions, with 4.6% of cases showing double aneuploidy and only 0.4% showing 3 or more aneuploidies (2).

The high rate of complex aneuploidy in cleavage and blastocyst stage embryos even among young patients suggests multiple mitotic errors in the first few cell divisions, which would likely lead to developmental arrest (2). Therefore, if transferred, such embryos would be expected not to implant or to miscarry. Historically, embryos with multiple chromosomal abnormalities have therefore been de-selected for transfer or even discarded. However, recently Lin et al. reported a healthy live birth following chaotic embryo transfer (3), calling into question the assumed non-viability of chaotic embryos. Might some of these embryos correct multiple aneuploidies and become euploid? It is plausible that any euploid population of cells could have a higher survival rate and a higher mitotic rate, and if abnormal cells undergo apoptosis, a euploid embryo could result. This could explain the low rate of complex aneuploidy seen in miscarriages. An additional explanation is that imperfections in the biopsy, amplification, and/or NGS PGT-A process occasionally lead to noisy reads, that are interpreted as multiple chromosomal abnormalities, but actually reflect artifact. For such embryos, re- testing may result in euploid results.

Small studies (published in abstract form only) have evaluated the reproducibility of chaotic results from NGS-based PGT-A. A retrospective cohort study evaluated 58 'chaotic' embryos via PGT-A of re-biopsy samples. Thirty-eight percent (n=22) of embryos had euploid re-biopsy results (4). Our group reported re-biopsy of 64 embryos initially classified as chaotic and identified 17% (n=11) of embryos in the cohort as euploid and only 67% concordance between initial and re-biopsy sample results (5). Four blastocysts with euploid results on re- biopsy were transferred, resulting in two ongoing pregnancies. Furthermore, we have pooled data from multiple IVF clinics within our network that have conducted re-biopsy of embryos with multiple aneuploidies and found that overall, 22% had euploid PGT-A results on re-biopsy (Background Table, unpublished data).

In anticipation of conducting a prospective observational study to characterize the nature of PGT-A results indicating 3 or more aneuploidies, we have begun to catalog and hold these embryos in storage. To date, 112 patients with have explicitly expressed interest in contributing 128 embryos resulted as 'chaotic' or 'complex aneuploid' of 3-5 chromosomes, for the purposes of this research, and we anticipate identifying multiples of this number upon a

retrospective database search and with prospective accumulation of additional PGT-A results. Following a retrospective database search, we have identified a total of 274 'chaotic' and 5251 'complex aneuploid' embryos having been reported using NGS based PGT-A. Limited data exist on the reproductive potential of embryos classified as having multiple chromosomal abnormalities, and preliminary data, including from our center, suggest a high false positive rate. The large volume of ART performed within our network represents a unique opportunity to characterize the clinical significance of these results, in the hopes of minimizing embryo wastage and maximizing live birth from IVF cycles using PGT-A.

The aim of this study is to evaluate the reproductive potential of embryos classified as "complex aneuploid" of three or more chromosomes or "chaotic" on initial trophectoderm biopsy sample analyzed by next generation sequencing based preimplantation genetic testing for aneuploidy. We plan to do this by prospectively enrolling patients with embryos classified as such, re-biopsy of the embryos, and analysis of repeat biopsy samples. We also plan to have an independent, blinded geneticist make diagnoses, as possible, based on the NGS profiles.

ELIGIBILITY:
Inclusion Criteria:

* Having ≥ 1 embryo classified as whole chromosome chaotic or complex aneuploid of 3 or more chromosomes following preimplantation genetic testing for aneuploidy using an NGS based platform Signed informed consent

Exclusion Criteria:

* Embryos not meeting complex/chaotic criteria Patients declining consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with one or more embryos in storage that meet criteria for Chaotic or Complex Aneuploidy by PGT-A with NGS
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Reproducibility | one year
  To evaluate embryos with 3 or more chromosomes deemed aneuploid with NGS-based PGT-A by performing repeat biopsy and analyzing with NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Devine, MD, Study Director — Shady Grove Fertility; Benjamin S Harris, MD, MPH, Principal Investigator — Shady Grove Fertility
Locations (11):
- United States (10):
  - IVF Florida Reproductive Associates, Margate, Florida
  - Shady Grove Fertility, Atlanta, Georgia
  - Fertility Center of Illinois, Highland Park, Illinois
  - Shady Grove Fertility, Rockville, Maryland
  - Shady Grove Fertility, Towson, Maryland
  - Shady Grove Fertility, Cary, North Carolina
  - Shady Grove Fertility, Chesterbrook, Pennsylvania
  - Shady Grove Fertility, Fairfax, Virginia
  - Shady Grove Fertility, Norfolk, Virginia
  - Shady Grove Fertility, Richmond, Virginia
- SGFertility Chile Medicina Reproductiva, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided